CLINICAL TRIAL: NCT05163665
Title: Cost-effective Analysis of Two Approximation Devices in Closure of Gastrointestinal Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Salmaan Azam Jawaid, MD, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-50701
Record Dates: First submitted 2021-12-01; First posted 2021-12-20 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Gastrointestinal Neoplasms
Keywords: Closure of GI defects
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Through-the-Scope clip group (Experimental): Through the scope Dual Action Tissue Clip (DAT) clipping equipment and technique performed in closure of GI defect area after polyp removal.
  Interventions: Procedure: Closure type
- X-Tack suturing group (Active Comparator): Use of Endoscopic Helix Tacking System (X-Tack) by Apollo Endosurgery for the closure of GI defect after polyp removal.
  Interventions: Procedure: Closure type

INTERVENTIONS:
Procedure: Closure type — Patients will have their endoscopic submucosal dissection (ESD) or endoscopic mucosal resection (EMR) as per standard-of-care. Afterwards, patient will receive one of two intervention options for the closure of the GI defect following polyp removal.

SUMMARY:
This is a prospective, randomized research trial that aims to evaluate the clinical results of two different approximation methods to close the tissue defect caused by removing gastrointestinal polyps.

DETAILED DESCRIPTION:
Closure of GI defects after endoscopic resection decreases the rate of post resection bleeding. Traditionally, standard TTS clips have been used to close GI wall defects with some success. However, complete apposition of the resection wall edges occurs only 68% of the time. Endoscopic suturing with the traditional Overstitch device can achieve complete closure in almost 100% of defects. However, this device is costly, requires the use of a double channel therapeutic endoscope, and at times can be difficult to maneuver. Recently, a novel FDA approved TTS tissue helix and suture device (X-tack) was developed to overcome the challenges of the traditional Overstitch device. Animal models have demonstrated the X-tack system is superior to TTS in effecting large mucosal defects and maintain similar durability. At BCM, we have been using the X-tack system routinely in closure of GI defects.

ELIGIBILITY:
Inclusion Criteria:

* Patient is greater than or equal to 18 years of age.
* Patient can provide informed consent.
* Patient is referred for endoscopic mucosal resection (EMR) or endoscopic submucosal dissection (ESD) of gastric, small bowel, or colorectal lesion.
* Post resection defect > 3cm.
* Lesion 2cm or greater from the dentate line.

Exclusion Criteria:

* Patient is < 18 years of age.
* Patient refused and/or unable to provide consent.
* Patient is pregnant.
* Patient is currently incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
Cost of each closure | Day 1
  Total cost amount for equipment used in closure of GI defect

SECONDARY OUTCOMES:
Rate of complete closure of GI defect | Day 1 (end of procedure)
  Complete closure achieved by assigned closure type as assessed by performing physician
Successful Tissue approximation | Day 1 (End of procedure)
  Less than or equal to 15mm of visible resection bed at its widest portion after the device is used for tissue approximation

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Derived] Jawaid S, Khalaf M, Ayoub F, Zabad N, Fikry A, Daba G, Mercado M, Keihanian T, Othman M. RCT comparing the clinical efficacy and costs of two tissue approximation devices in the closure of large post-endoscopic resection defects. Surg Endosc. 2025 Aug;39(8):5442-5453. doi: 10.1007/s00464-025-11876-1. Epub 2025 Jul 10. PMID 40640617